CLINICAL TRIAL: NCT02023957
Title: Interactive Computer-assisted Screening for Mental Health in Primary Care
Brief Title: A Pilot With Interactive Computer-assisted Screening for Mental Health in Primary Care
Acronym: iCAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: York University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); North York General Hospital (Other)
Responsible Party: Principal Investigator, Farah Ahmad, Associate Professor, York University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: e2013 - 291
Record Dates: First submitted 2013-12-12; First posted 2013-12-30 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-06

CONDITIONS: Mental Health Disorders
Keywords: Interactive Health-risk assessment; Primary Care; Randomized; Open Label; Efficacy Study

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interactive computer-assisted screening (Experimental): Eligible patients completed the interactive computer-assisted screening (iCAS) tool in English or Spanish before seeing the consenting clinician. Participating patients then received the iCAS generated tailored recommendation sheet. Participating clinicians received the iCAS generated risk report.
  Interventions: Behavioral: Interactive computer-assisted screening (iCAS)
- Usual Care (No Intervention): Eligible patients randomized to the control group completed their standard visit to the participating clinician. There was no pre-visit health risk screening. There were no tailored reports for the patients or clinicians.

INTERVENTIONS:
Behavioral: Interactive computer-assisted screening (iCAS)
  Arms: Interactive computer-assisted screening

SUMMARY:
The current protocol pertains to the evaluation of the interactive computer-assisted screening (iCAS) tool through a pilot randomized control trial. The purpose of this evaluation is to determine the efficacy of the iCAS tool in improving clinician's detection of common mental health conditions (i.e. major depression/generalized anxiety/post-traumatic stress disorder/alcohol dependence), and patients' discussion on mental health.

DETAILED DESCRIPTION:
The iCAS tool is a health-risk assessment survey that is completed by adult patients using touch-screen iPad device in their waiting time before seeing their clinician (family physician or nurse practitioner). The computer program generates tailored risk-report for the clinician and a simple recommendation sheet for the patient, with community resources and health information, at the point of care. The iCAS tool currently includes validated screening scales for depression, generalized anxiety, posttraumatic stress disorder and alcohol abuse. There are some questions on the social determinants of mental health as well. The current versions of the tool are in English and Spanish; a Chinese language version will also be developed.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Speak/read Spanish
* Speak/read English
* Visiting the consenting clinician

Exclusion Criteria:

* Patient accompanied by a family member for interpretation
* New patients coming for first visit
* Patients feeling unwell (self-report)
* Inability of the research staff to offer study details in privacy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2013-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Clinician Detection (probable, sub-clinical, confirmed) of major depression or generalized anxiety or post-traumatic stress disorder or alcohol dependence | Day 1
  Chart review for the index visit
Patient discussion on mental health | Day 1
  Exit Survey of patients after the index visit

SECONDARY OUTCOMES:
Patient intention to see a mental health counselor | Day 1
  Exit Survey of patients after the index visit
Patient satisfaction with health services | Day 1
  Exit Survey of patients after the index visit
Patient enablement to cope with these conditions | Day 1
  Exit Survey of patients after the index visit
Patient adherence to follow-up advice and referrals to mental health support | 3 month
  Chart review

OTHER OUTCOMES:
Symptom reduction | 6 month
  Measurement of this outcome depends on availability of funds for follow-up phone interviews

CONTACTS AND LOCATIONS:
Overall Officials: Farah Ahmad, PhD, Principal Investigator — York University
Locations (1):
- York University, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ahmad F, Lou W, Shakya Y, Ginsburg L, Ng PT, Rashid M, Dinca-Panaitescu S, Ledwos C, McKenzie K. Preconsult interactive computer-assisted client assessment survey for common mental disorders in a community health centre: a randomized controlled trial. CMAJ Open. 2017 Mar 1;5(1):E190-E197. doi: 10.9778/cmajo.20160118. eCollection 2017 Jan-Mar. PMID 28401134
- [Derived] Ferrari M, Ahmad F, Shakya Y, Ledwos C, McKenzie K. Computer-assisted client assessment survey for mental health: patient and health provider perspectives. BMC Health Serv Res. 2016 Sep 23;16(1):516. doi: 10.1186/s12913-016-1756-0. PMID 27663508